CLINICAL TRIAL: NCT03833921
Title: Evaluation of Response to Abiraterone/Prednisone by Race/Ethnicity, PSA Decline and Genetic Variation in Proteins Involved in Androgen Metabolism in Metastatic Hormone Naive Prostate Cancer
Brief Title: Evaluation of Response to Abiraterone/Prednisone by Race/Ethnicity and Other Factors in Metastatic Hormone Naive Prostate Cancer
Acronym: APRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Martha Mims (Other)
Responsible Party: Sponsor-Investigator, Martha Mims, Professor, Medicine - Hematology and Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-44335
Record Dates: First submitted 2019-02-01; First posted 2019-02-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer
Keywords: Abiraterone acetate; hormone naive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abiraterone acetate + prednisone (Other): All subjects will receive abiraterone acetate and prednisone, as per standard of care. Abiraterone acetate will be administered orally as 1000 mg once daily along with 5 mg of oral prednisone twice per day. Subjects will continue to take abiraterone acetate and prednisone until confirmed disease progression.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg orally daily until disease progression
  Other Names: Zytiga
Drug: Prednisone — 5 mg oral low dose prednisone, twice daily

SUMMARY:
The investigators are conducting this study with men that have prostate cancer and are getting standard of care treatment with the drugs abiraterone acetate and prednisone. The study will follow men with prostate cancer from initiation of participation in the study and for up to 10 years. The reason for the study is that researchers think that there may be a connection between the race and ethnicity of men with prostate cancer and how well the standard treatments work for the participants.

DETAILED DESCRIPTION:
This is a single arm study in metastatic hormone naïve prostate cancer. Standard of care in these men is either to offer Androgen deprivation therapy (ADT) + abiraterone acetate/low-dose prednisone or, in men with higher tumor burden, to offer ADT + Docetaxel/prednisone. The investigator's experience is that even men with increased tumor burden often opt for abiraterone because of the improved side effect protocol as compared to chemotherapy.

Approximately 130 PSA response evaluable subjects will be enrolled, of which the investigators expect 50% to be African American based on clinic population and previous experience with clinical trial enrollment.

The study will enroll men with newly diagnosed hormone naïve prostate cancer within 42 days of receiving the first dose of ADT (LHRH agonist or antagonist) or undergoing orchiectomy. Patients will continue ADT throughout the study. Abiraterone acetate and low dose prednisone will continue until progression as defined by standard PCWG2 criteria.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologically or cytologically proven diagnosis of adenocarcinoma of the prostate. All patients must have metastatic disease as evidenced by soft tissue and/or bony metastases prior to initiation of androgen deprivation therapy (ADT). NOTE: ADT does not include treatment with anti-androgens such as bicalutamide or flutamide or five alpha reductase inhibitors such as finasteride or dutasteride.
* Patients must have radiographic assessments of all disease including bone scan (or PET scan) within 42 days prior to registration. All disease will be assessed and documented on the appropriate CRF.
* Patients must have had no more than 42 days of prior castration (medical or surgical) for metastatic prostate cancer prior to starting abiraterone. The start date of medical castration is considered the day the patient first received an injection of a LHRH agonist/antagonist (or orchiectomy), not an oral antiandrogen. • If the method of castration was luteinizing hormone releasing hormone (LHRH) agonist or antagonist (i.e., leuprolide, goserelin or degarelix), the patient must be willing to continue the use of LHRH agonist/antagonist and add Abiraterone + Prednisone treatment. • If the patient was on an antiandrogen (e.g. bicalutamide, flutamide), the patient must be willing to switch over to Abiraterone + Prednisone treatment. There is no limit on how many days a patient may have been on an antiandrogen (e.g. bicalutamide, flutamide) or a five alpha reductase inhibitor (e.g. finasteride or dutasteride) prior to going on study and no washout is required.
* Patients may have received prior ADT - neoadjuvant and/or adjuvant setting only - but it must not have lasted for more than 36 months. Single or combination therapy allowed. At least 6 months must have elapsed since completion of ADT in the neoadjuvant and/or adjuvant setting, and serum testosterone must be > 50 ng/dL (non-castrate levels) within 28 days prior to registration. NOTE: Serum testosterone assessment is required for eligibility for only those patients with prior treatment with neoadjuvant or adjuvant ADT.
* Patients who are deemed to have high-risk or extensive metastatic, hormone sensitive prostate cancer (mHSPC) per "clinical judgment" of the treating physician are eligible for enrollment if the participants are unsuitable candidates for docetaxel or if the participants have declined docetaxel therapy.
* Patients may have received prior surgery. For all major surgeries, at least 14 days must have elapsed since completion and patient must have recovered from all major side effects of surgery per investigator's assessment.
* Patients may have received or plan to receive concurrent bone targeting agents that do not have an effect on PSA (e.g. denosumab or bisphosphonate).
* Patients must have no plans to receive any other experimental therapy while on the protocol treatment. Previous experimental therapy must have been completed at least 28 days prior to registration.
* Patients must have a complete physical examination and medical history within 28 days prior to registration.
* Patients must have a PSA ≥ 10 ng/mL obtained within 90 days prior to registration.
* Patients must have a QTc interval < 461 msec on the 12 lead ECG within 42 days prior to registration. Patients with asymptomatic or incidental bundle branch blocks may have QTc measured by a cardiologist or standard formulas such as Bazett's or Fridericia's to adjust for pre-existing blocks.
* Patients must have adequate hepatic function, within 28 days prior to registration, as evidenced by: • bilirubin ≤ 2 x institutional upper limit of normal (ULN), and • SGOT (AST) and SGPT (ALT) ≤ 3 x institutional ULN, or ≤ 5 x institutional ULN if liver metastases are present.
* Patients must have adequate renal function, within 28 days prior to registration, as evidenced by calculated creatinine clearance ≥ 40 mL/min using a serum creatinine or by 24-hour urine creatinine (using Cockroft-Gault equation).
* Patients must have adequate hematologic function, within 28 days prior to registration as evidenced by:

  * leukocytes ≥ 3,000/mcL,
  * absolute neutrophil count (ANC) ≥ 1,500/mcL,
  * hemoglobin ≥ 9 g/dL, and
  * platelets ≥ 100,000/mcL.
* Patients must have a Zubrod performance status of 0-2. Zubrod performance status 3 will be allowed if from bone pain only.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
* Patients must be ≥ 18 years of age.
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Voluntary written informed consent must be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients with known brain metastases are not eligible. Brain imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms suggestive of brain metastasis. But, if brain imaging studies are performed, patients must be negative for disease.
* Patients must not have received prior and/or must not have any plans for receiving concomitant therapy with ketoconazole, aminoglutethimide, or enzalutamide (MDV3100). Concurrent megestrol for hot flashes is allowed.
* Patients must not have received any prior cytotoxic chemotherapy for metastatic prostate cancer. Prior cytotoxic chemotherapy with curative intent in the neoadjuvant or adjuvant setting is allowed. At least 2 years must have elapsed since completion of cytotoxic chemotherapy in the neoadjuvant and/or adjuvant setting.
* Patients must not have New York Heart Association Class III or IV heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction, or serious uncontrolled cardiac arrhythmia within 6 months prior to registration. (Note: Androgen deprivation therapy may prolong the QT/QTc interval. Patients with congenital long AT syndrome, congestive heart failure, frequent electrolyte abnormalities, and patients taking drugs known to prolong the QT interval may be at increased risk.)
* Patients with a known history of primary and secondary adrenal insufficiency are not eligible.
* Patients must not be known to have hypersensitivity to abiraterone or to LHRH agonist/antagonist.
* Patients must not have known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of abiraterone, including difficulty swallowing oral medications per investigator's clinical judgement.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2038-04 (Estimated)

PRIMARY OUTCOMES:
PSA Response Rate | Treatment start until 7 months after start of ADT
  The proportion of subjects with PSA levels less than 4 ng/ml at the given time point.

SECONDARY OUTCOMES:
Depth of PSA Response | Treatment start until nadir, or up to 7 months after start of ADT if no nadir
  Measure of the absolute amount of change in PSA levels, or measure of proportional change in PSA levels.
Frequency of Potentially Deleterious Polymorphisms | Measured at baseline
  Number of potentially deleterious polymorphisms in proteins involved in androgen metabolism, stratified by race/ethnicity.
Progression Free Survival | Treatment start until event or up to 3 years after start of ADT
  Measure of time until disease progression.
Time to PSA Progression | Treatment start until event or up to 3 years after start of ADT
  Measure of time until PSA progression.
Time to Subsequent Prostate Cancer Therapy | Treatment start until event or up to 3 years after start of ADT
  Measure of time until start of subsequent prostate cancer therapy.
Time to Initiation of Chemotherapy | Treatment start until event or up to 3 years after start of ADT
  Measure of time until start of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Mims, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Ben Taub General Hospital, Houston, Texas
  - Dan L. Duncan Comprehensive Cancer Center at Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.